CLINICAL TRIAL: NCT00523978
Title: A Randomized, Controlled Clinical Trial of Catheter Cryoablation in the Treatment of Paroxysmal Atrial Fibrillation.
Brief Title: A Clinical Study of the Arctic Front Cryoablation Balloon for the Treatment of Paroxysmal Atrial Fibrillation
Acronym: Stop-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS-023
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Flecainide; Sotalol; Propafenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Experimental subjects received cryoablation intended to isolate the pulmonary veins and ablate arrhythmia foci. If necessary, experimental subjects were allowed a previously failed Study Atrial Fibrillation Drug (AF Drug).
  Interventions: Device: Arctic Front® Cryoablation Catheter
- Control (Active Comparator): Control Subjects were treated with an AF Drug (flecainide, propafenone, or sotalol) that they had not previously failed.
  Interventions: Drug: Flecainide or Sotalol or Propafenone

INTERVENTIONS:
Device: Arctic Front® Cryoablation Catheter — Experimental Subjects received cryoablation intended to isolate the pulmonary veins and ablate arrhythmia foci with the cryoablation catheter system.
  Other Names: Arctic Front® Cardiac CryoAblation Catheter System; Artic Front®
  Arms: Experimental
Drug: Flecainide or Sotalol or Propafenone — Flecainide 200 mg / day Propafenone 450 mg / day Propafenone-SR 650 mg / day Sotalol 240 mg / day
  Other Names: Tambocor; Sotalol; Propafenone
  Arms: Control

SUMMARY:
This study (STOP AF) is a prospective, randomized, controlled, multicenter, pivotal clinical investigation conducted at 26 investigational sites in the United States and Canada. Subjects with paroxysmal atrial fibrillation (PAF) referred for ablative intervention after efficacy failure of one or more Study Atrial Fibrillation (AF) Drugs (flecainide, propafenone or sotalol) were randomized 2:1 to cryoablation intervention (Experimental Subjects, ES) or to a Study AF Drug (Control Subjects, CS). Subjects were followed for 12 months with scheduled and symptom-driven assessments to detect recurrent atrial fibrillation by means of periodic electrocardiograms, weekly scheduled trans-telephonic monitoring, patient-initiated trans-telephonic monitoring, and 24-hour Holter monitoring at 6 and 12 months. The first 90 days after study therapy was initiated was considered a blanked period for all subjects.

DETAILED DESCRIPTION:
STOP AF (PS-023) is a randomized, controlled study of subjects 18 to 75 years old who had been referred for ablative intervention after failing one or two (but not all three) anti-arrhythmic drugs used in the treatment of AF (flecainide, propafenone and sotalol). Study subjects were randomized into two arms: the cryoablation (treatment) arm and the membrane-active antiarrhythmic drug (control) arm. A 90- day blanked follow-up period, including reablation and medication adjustments was applied in both arms to optimize therapies. All subjects underwent follow-up assessments at 1, 3, 6, 9 and 12 months, weekly transtelephonic monitoring, 24-hour Holter monitoring and CT/MRI of the pulmonary veins(at 6 and 12 months) during the trial period. Control subjects who were confirmed to be chronic treatment failures were permitted to crossover to cryoablation in this trial.

Acute procedural success was defined for subjects that underwent cryoablation and demonstrated electrical isolation in ≥ 3 Pulmonary Veins (PVs) at the conclusion of the first protocol-defined cryoablation procedure using the Arctic Front® Cardiac CryoAblation Catheter System.

The primary effectiveness endpoint was defined as having acute procedural success and freedom from chronic treatment failure (CTF) for experimental subjects, and freedom from CTF for control subjects. Freedom from (CTF) was defined for both groups as the occurrence of detectable AF during a non-blanked follow-up period, or an AF Intervention, or the use of a non-study AF drug at any time.

The co-primary safety outcome measures were Cryoablation Procedure Events (CPEs) in cryoablated subjects and Major Atrial Fibrillation Events (MAFEs) in both groups. CPEs were device- or procedure-related serious adverse events.

Other safety assessments were made during the course of the STOP AF trial specific to pulmonary vein stenosis (PVS) and phrenic nerve injury.

ELIGIBILITY:
Inclusion Criteria:

* Documented Paroxysmal Atrial Fibrillation (PAF): PAF diagnosis, 2 episodes of PAF within the last 2 months, at least 1 episode of PAF must be documented
* Age 18-75
* Documented Effectiveness Failure of one (1) AF drug
* Willing to be randomized to either group and do full 12 month follow-up
* Able to follow standardized AF drug protocol

Exclusion Criteria:

* Any cardioversion within 3 months or more than 2 within 2 years
* Amiodarone within 6 months
* LA size > 5.0cm
* Previous LA ablation/surgery, structural heart disease, heart failure class III or IV
* Hypertrophic cardiomyopathy, Mitral prosthesis
* Unstable angina, uncontrolled hyperthyroidism
* Stroke or TIA within 6 months, MI within 2 months, cardiac surgery within 3 months
* Thrombocytosis, thrombocytopenia
* Any condition contraindicating chronic anticoagulation
* EF <40%
* Pregnancy
* Life expectancy <1year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-10; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L. Packer, MD, Principal Investigator — Mayo Clinic
Locations (26):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Cedar Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford Hospital, Stanford, California
  - Colorado Cardiac Alliance -- Memorial Hospital, Colorado Springs, Colorado
  - Mayo Clinic- Jacksonville, Jacksonville, Florida
  - BayHeart Group -- St-Joseph's Hospital, Tampa, Florida
  - Emery Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Iowa Heart Center, Des Moines, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Health, Philadelphia, Pennsylvania
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Inova Research Center, Falls Church, Virginia
  - Sentara CV Research Institute, Norfolk, Virginia
  - Medical College of Virginia, Richmond, Virginia
  - Cardiology Associates of Green Bay, Green Bay, Wisconsin
  - Arrhythmia Center of Southern WI, Milwaukee, Wisconsin
- Canada (3):
  - London Medical Health Sciences, London, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Laval Hospital, Ste-Foy, Quebec

REFERENCES:
- [Derived] Packer DL, Kowal RC, Wheelan KR, Irwin JM, Champagne J, Guerra PG, Dubuc M, Reddy V, Nelson L, Holcomb RG, Lehmann JW, Ruskin JN; STOP AF Cryoablation Investigators. Cryoballoon ablation of pulmonary veins for paroxysmal atrial fibrillation: first results of the North American Arctic Front (STOP AF) pivotal trial. J Am Coll Cardiol. 2013 Apr 23;61(16):1713-23. doi: 10.1016/j.jacc.2012.11.064. Epub 2013 Mar 21. PMID 23500312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators at 26 sites in the United States and Canada, enrolled and randomized a total of 245 study subjects, during the 21 months trial period, between 10 October 2006 and 30 June 2008.
Groups:
- Cryoablation: an experimental group receiving cryoablation and, optionally, a previously failed Atrial Fibrillation Drug.3 Subjects withdrew consent 5 subjects were a screen failure. Therefore N=163 for Experimental group.
- Standard Treatment With Drugs Only: a control group receiving only an Atrial Fibrillation Drug. 4 Subject withdrew consent and 1 subject was a screen failure. Therefore- Control Treatment group N= 82.
Period: Overall Study
Arm/Group | Cryoablation | Standard Treatment With Drugs Only
Started | 171 | 87
Completed | 162 | 79
Not Completed | 9 | 8
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Screen Failures | 5 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoablation | Standard Treatment With Drugs Only | Total
Number analyzed (Participants) | 163 | 82 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (0.73) | 56.4 (1.04) | 56.6 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 18 | 56
  Male | 125 | 64 | 189
Region of Enrollment [Number; unit: participants]
  United States | 123 | 63 | 186
  Canada | 40 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Acute Procedural Success (APS)
Description: Acute Procedural Success was defined as a demonstration of electrical isolation in ≥ 3 Pulmonary Veins (PVs) at the conclusion of the first protocol-defined cryoablation procedure. APS was decided at the end of the procedure the mean time was calculated for the time frame.
Time Frame: 371.4 Minutes (Average)
Population: Subjects evaluated were from the modified Intent to Treat subset (mITT)or subjects that were enrolled, randomized and received treatment.
Measure: Number; unit: participants
Groups:
- Cryoablation: Experimental group or group that were cryoablated with Arctic Front® Cardiac CryoAblation Catheter System, including the FlexCath® Steerable Sheath and Freezor® MAX Cardiac Cryoablation Catheter
Arm/Group | Cryoablation
Number analyzed (Participants) | 163
participants | 160

2. Primary Outcome: Freedom From Chronic Treatment Failure (CTF)
Description: Subjects that did not have or were free of CTF. CTF was defined as the occurence of an Atrial Fibrillation (AF) intervention, use of non-study AF drug therapy, or the occurence of detectable AF which is is defined as an episode of AF, documented in a tracing, and lasting more than 30 seconds, occurring during a Non Blanked Follow-up Period.
Time Frame: 12 month follow up period
Population: This section includes data for subjects who were randomized, received treatment and were followed through 12-Months post randomized treatment regardless of AF Drug usage. Subjects who experienced Acute Procedural Failure in the Experimental group were not included in this analysis of post-procedural failure causes.
Measure: Number; unit: participants
Groups:
- Cryoablation: Experimental group or subjects that were cryoablated with Arctic Front® Cardiac CryoAblation Catheter System, including the FlexCath® Steerable Sheath and Freezor® MAX Cardiac Cryoablation Catheter
- Standard Treatment With Drugs Only: A control group receiving only an Atrial Fibrillation Drug who have not previously failed a AF study drug.
Arm/Group | Cryoablation | Standard Treatment With Drugs Only
Number analyzed (Participants) | 163 | 82
participants | 117 | 6

3. Primary Outcome: Treatment Success
Description: Treatment Success was defined as Acute Procedure Success (APS) and freedom from Chronic Treatment Failure (CTF) for Experimental Subjects, and freedom from CTF for Control Subjects. Under this pre-specified definition of Treatment Success, Experimental Subjects must have had APS and remained free of CTF during the 12-month follow-up duration, while Control Subjects must have remained free of CTF during the 12-month follow-up duration.
Time Frame: 12 months
Population: The mITT population consisted of all subjects, who were enrolled, randomized and received treatment
Measure: Number; unit: participants
Arm/Group | Cryoablation | Standard Treatment With Drugs Only
Number analyzed (Participants) | 163 | 82
participants | 114 [62.3 to 76.9] | 6 [2.7 to 15.2]
Statistical Analysis 1: Comparison: Cryoablation vs Standard Treatment With Drugs Only; The null hypothesis is the success rate in experimental group is less than and equal to the one in control group. This comparison of the rates was performed using a 2-sided Fisher's Exact. A sample size of 240(160 experimental and 80 control) is required to provide 80% power to detect the treatment difference using a 2-sided (alpha = 0.05)Fisher's Exact Test of binomial proportions assuming the success rate was 40% for control and 60% for treatment; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Primary Outcome: Freedom From Major Atrial Fibrillation Events (MAFEs)
Description: Subjects that did not have or were free of MAFEs. MAFEs were serious adverse events categorized as cardiovascular death, myocardial infarction, stroke, or hospitalization for AF recurrence/ablation, flutter ablation, embolic events, heart failure, hemorrhage or anti-arrhythmic drug treatment.
Time Frame: 12 Months
Population: mITT set included all subjects (82 CS, 163 ES) who were enrolled, randomized, and received treatment.
Measure: Number; unit: participants
Arm/Group | Cryoablation | Standard Treatment With Drugs Only
Number analyzed (Participants) | 163 | 82
participants | 158 | 75
Statistical Analysis 1: Comparison: Cryoablation vs Standard Treatment With Drugs Only; The null hypothesis is the proportion of subjects free from MAFE in the experimental group is inferior to that in the control group using 10% non-inferiority margin.A sample size of 160 evaluable cryoablation and 80 control subjects (one-sided α = 0.05, 2:1 randomization) was required to provide 80% power assuming the rate of free from MAFE at 12 months 80.5 and 77% in experimental and control groups respectively; Test type: Non-Inferiority or Equivalence — A non-inferiority margin was selected based on literature review; p < 0.001, t-test, 1 sided

5. Primary Outcome: Cryoablation Procedure Events (CPEs)
Description: Subjects that had CPEs. CPEs were device- or procedure-related serious adverse events (SAE) categorized as access site complications, cardiac damage, pulmonary vein (PV) stenosis, embolic complications, arrhythmias, unresolved phrenic nerve palsy and death.
Time Frame: To end of ablation procedure
Population: Data for subjects who were randomized to the Experimental group and received cryoablation therapy were included in this analysis. All CPEs reported in the Experimental group were included in the analysis regardless of their association with the first or a repeat cryoablation.
Measure: Number; unit: participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 163
participants | 5
Statistical Analysis 1: Comparison: Cryoablation; The test hypothesis is UCBExperimental_CPE ≥ 14.8% vs UCBExperimental_CPE < 14.8%.The performance goal 14.8% was chosen based on a review of SSEDs for similar types of ablation trials.The expected rate for CPEs in a well-monitored trial of left atrial RF ablation for AF was estimated to be 10% (corresponding to a CPE-free rate of 90%).In a trial with 160 subject, the resulting one-sided 95% upper confidence bound would be 14.8%; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: All pharmacologic and ablative treatments and arrhythmic disease adverse events on study subjects were followed through 12 months of follow-up.
Description: All serious adverse events (SAE) were adjudicated by the CEC to the protocol definitions.
Arm/Group | Cryoablation | Standard Treatment With Drugs Only
Serious Adverse Events (participants affected / at risk) | 20/163 | 12/82
Other Adverse Events (participants affected / at risk) | 19/163 | 16/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation (N=163) | Standard Treatment With Drugs Only (N=82)
A fib persistent-drug load (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal wall hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute pyelonephritis 2º to vesical catheter (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute renal failure requiring dialysis (Renal and urinary disorders) | 0 (0) | 1 (1)
Altered mental status S/P cardiac arrest (Psychiatric disorders) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter-recurrent (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary arrest with resuscitation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary decompensation-etiology uncertain (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Escherichia coli bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Focal hemorrhage of ileum 2º to warfarin induced coagulopathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematoma from left groin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increasing persistent A fib (Cardiac disorders) | 0 (0) | 1 (1)
Interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Left atrial appendage thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Left popliteal deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Left upper + lower pulmonary vein stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Multiple organ failure (General disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Non Q wave myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Non bacterial meningitis (Nervous system disorders) | 0 (0) | 1 (1)
Occlusion left inferior pulmonary vein (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (tamponade) (Cardiac disorders) | 1 (1) | 0 (0)
Persistent atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Physical deconditioning 2º to procedural complications and immobilization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonia left lower lobe (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolus (Vascular disorders) | 1 (1) | 0 (0)
Rapid atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Recurrent atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Recurrent rapid A fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Right diaphragm paresis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right lung blebs with persistent air leak (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right wrist heparin lock insertion site infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis induced hypotension (Infections and infestations) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Subdural hematoma from fall (Vascular disorders) | 0 (0) | 1 (1)
Wegener's granulomatosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Worsened AF with rapid ventricular response (Cardiac disorders) | 1 (1) | 0 (0)
Worsening AF (Cardiac disorders) | 2 (2) | 1 (1) — Worsening Atrial Fibrillation
Worsening atrial flutter (Cardiac disorders) | 1 (1) | 1 (2)
Worsening atrial fib-flutter (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation (N=163) | Standard Treatment With Drugs Only (N=65)
Atrial Fibrillation (Cardiac disorders) | 14 (14) | 16 (16)
Atrial Flutter (Cardiac disorders) | 18 (18) | 10 (10)
Bradycardia (Cardiac disorders) | 0 (0) | 4 (4)
Fatigue (General disorders) | 12 (12) | 9 (9)
Chest Pain (General disorders) | 9 (9) | 4 (4)
Chest Discomfort (General disorders) | 4 (4) | 8 (8)
Asthenia (General disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 17 (17) | 11 (11)
Dizziness (Nervous system disorders) | 15 (15) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Nausea (Gastrointestinal disorders) | 9 (9) | 9 (9)
Bronchitis (Infections and infestations) | 10 (10) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Hypertension (Vascular disorders) | 6 (6) | 4 (4)
Hypotension (Vascular disorders) | 3 (3) | 5 (5)
international Normalised Ratio Increased (Investigations) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less